CLINICAL TRIAL: NCT04344405
Title: Vitamin D as a Key Player in Rheumatoid Arthritis Immune Response
Brief Title: Vitamin D as a Key Player in Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vit D in RA
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: the Immunomodulatory Effect
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vit D (Experimental)
  Interventions: Drug: Vitamin D
- control (Active Comparator)
  Interventions: Drug: Steroid Drug

INTERVENTIONS:
Drug: Vitamin D — vitamin D supplementation
  Arms: Vit D
Drug: Steroid Drug — control
  Arms: control

SUMMARY:
Rheumatoid arthritis (RA) is a systemic, chronic and inflammatory disease of joints linked to autoimmunity. Vitamin D was found to modulate cell growth, function of immune cells and anti-inflammatory action. The aim of this study was to investigate serum vitamin D level and some cytokines and to identify the correlation between vitamin D and these cytokines in RA.

Methods: Totally 60 RA patients without vitamin D supplement were involved in this study. The serum level of vitamin D, interleukin-6 (IL-6), IL-10, IL-35, tumor necrosis factor α (TNF-α) and C-reactive protein (CRP) were measure in all patients by enzyme-linked immunosorbent assay (ELISA) then they will divided into 2 groups, group I receive vit. D supplementation and group II will receive placebo and follow up for 3 months.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic, chronic and inflammatory disease of joints linked to autoimmunity. Vitamin D was found to modulate cell growth, function of immune cells and anti-inflammatory action. The aim of this study was to investigate serum vitamin D level and some cytokines and to identify the correlation between vitamin D and these cytokines in RA.

Methods: Totally 60 RA patients without vitamin D supplement were involved in this study. The serum level of vitamin D, interleukin-6 (IL-6), IL-10, IL-35, tumor necrosis factor α (TNF-α) and C-reactive protein (CRP) were measure in all patients by enzyme-linked immunosorbent assay (ELISA) then they will divided into 2 groups, group I receive vit. D supplementation and group II will receive placebo and follow up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* RA patients

Exclusion Criteria:

* Patients with inflammatory bowel disease patients with any other autoimmune diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
disease activity score 28 | 3 months
  disease activity score

CONTACTS AND LOCATIONS:
Locations (1):
- Manal Hassanien, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided